CLINICAL TRIAL: NCT04377594
Title: Individually DEsigned Ablation of Low Voltage Areas in Patients With Persistent Atrial Fibrillation, a Randomized Controlled Multicenter Trial
Brief Title: Ablation of Fibrotic Areas in Patients With Persistent Atrial Fibrillation.
Acronym: IDEAL-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Jensen-Urstad, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200212IDEALAF
Record Dates: First submitted 2020-04-23; First posted 2020-05-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation; Low voltage
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Randomization 1:1
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary vein isolation plus substrate modification (Experimental): Pulmonary vein isolation plus ablation of low voltage areas in the left atrium
  Interventions: Procedure: Radio frequency ablation
- Pulmonary vein isolation (Active Comparator): Pulmonary vein isolation
  Interventions: Procedure: Radio frequency ablation

INTERVENTIONS:
Procedure: Radio frequency ablation — Two different radio frequency ablation procedures

SUMMARY:
Brief summary: The objective of this study is to compare two different ablation strategies in participants with persistent atrial fibrillation and fibrotic areas in the left atrium. The participant will be randomized to pulmonary vein isolation or pulmonary vein isolation plus ablation of fibrotic areas.

DETAILED DESCRIPTION:
Background:

Atrial fibrillation (AF) is the most common arrhythmia in clinical practice with a prevalence of 2-3 percent in the population. Catheter ablation performing pulmonary vein isolation (PVI) is an established treatment, which aim to eliminate triggers from the pulmonary veins. This treatment is successful in most patients with paroxysmal AF. In many patients, especially the patients with persistent AF, this treatment is not sufficiently to achieve freedom from arrhythmia and symptoms.

There are several studies showing that fibrosis in the left atrium (LA) is an independent factor to relapse in AF after PVI. The fibrotic areas can be detected by measuring the voltage in the left atrium and creating a voltage map. There are non-randomized studies that suggest better results regarding reduction of arrhythmia burden after ablating the low voltage areas (LVAs). This ablation strategy is commonly used in clinical praxis although there are no randomized studies in this field.

Aim:

The objective of this study is to compare two different ablation strategies in participants with persistent atrial fibrillation and fibrotic areas in the left atrium. The participant will be randomized to PVI versus PVI plus ablation of LVAs.

The primary endpoint is freedom of atrial arrhythmias after 1 to 2 ablation procedures within 6 months measured at 12 months after the first ablation procedure without antiarrhythmic drugs. Secondary endpoints will be atrial arrhythmia burden, health related quality of life measured by AFEQT score, and RAND 36 and periprocedural complications; death, stroke/ TIA, tamponade, atrio-esophageal fistula, and atrioventricular block.

Study design:

Randomized controlled multicenter trial. The study will be single blinded. All the participants will undergo PVI and the substrate map will be collected during atrial pacing. The patients with LVA will be randomized in a 1:1 fashion to; PVI plus ablation of LVA or PVI alone. Follow up visits will be at 3, 6, 12, 18 and 24 months. Before ablation and at every follow up visit the participants will fill in arrhythmia symptom specific questionnaires (AFEQT and ASTA) and questionnaire about quality of life (RAND 36). The participants will register arrhythmia with a heart monitoring system if symptoms of arrhythmia and two times daily during two weeks before every follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. ECG-documented persistent or long-standing persistent atrial fibrillation according to European Society of Cardiology (ESC) definition
2. Symptoms e. g. palpitations, dyspnea, tiredness that is due to the atrial fibrillation.
3. Suitable candidate for catheter ablation.
4. Tried one or more antiarrhythmic drugs or unwilling to try antiarrhythmic drugs
5. Age ≥18 years.

Exclusion Criteria:

1. LA dimension >55 mm as determined by an echocardiography within the previous year
2. Acute coronary syndrome or coronary artery bypass surgery within 12 weeks
3. Severe aortic or mitral valvular heart disease using the ESC guidelines
4. Congenital heart disease
5. Prior surgical or percutaneous AF ablation procedure or atrioventricular-nodal ablation
6. Medical condition likely to limit survival to < 1 year
7. New York Heart Association (NYHA) class IV heart failure symptoms
8. Contraindication to oral anticoagulation
9. Renal failure requiring dialysis
10. AF due to reversible cause
11. Pregnant and fertile women without anticonception
12. History of non-compliance to medical therapy
13. Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2026-04-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Freedom from Atrial Arrhythmia | From 3 months (blanking period) to 12 months after the first ablation procedure
  Freedom from documented atrial arrhythmias >30 seconds at 12 months after 1 or 2 ablation procedures within 6 months without antiarrhythmic drugs

SECONDARY OUTCOMES:
Number of Participants with Freedom from Atrial Arrhythmia after 1 Ablation Procedure without Antiarrhythmic Drugs (AAD) | From 3 months (blanking period) to 12 months after the first ablation procedure
  Freedom from documented atrial arrhythmias >30 seconds at 12 months after 1 ablation procedure without antiarrhythmic drugs
Number of Participants with Freedom from Atrial Arrhythmia after 1 Ablation Procedure with/ without AAD | From 3 months (blanking period) to 12 months after the first ablation procedure
  Freedom from documented atrial arrhythmias >30 seconds at 12 months after 1 ablation procedure with or without antiarrhythmic drugs
Number of Participants with Freedom from Atrial Arrhythmia after 1 or 2 Ablation Procedures with/ without AAD | From 3 months (blanking period) to 12 months after the first ablation procedure
  Freedom from documented atrial arrhythmias >30 seconds at 12 months after 1 or 2 ablation procedures with or without antiarrhythmic drugs
Number of Participants with Freedom from Atrial Fibrillation | From 3 months (blanking period) to 12 months after the first ablation procedure
  Freedom from documented atrial fibrillation >30 seconds at 12 months after 1 or 2 ablation procedures without antiarrhythmic drugs
Number of Participants with Freedom from Symptomatic Atrial Arrhythmias | From 3 months (blanking period) to 12 months after the first ablation procedure
  Freedom from documented symptomatic atrial arrhythmias >30 seconds at 12 months after 1 or 2 ablation procedures with or without antiarrhythmic drugs
Number of Participants with Freedom from Atrial Arrhythmias without AAD | From 3 months (blanking period) to 24 months after the first ablation procedure
  Freedom from documented atrial arrhythmias >30 seconds at 24 months after 1 or several ablation procedures without antiarrhythmic drugs
Number of Participants with Freedom from Atrial Arrhythmias with or without AAD | From 3 months (blanking period) to 24 months after the first ablation procedure
  Freedom from documented symptomatic atrial arrhythmias >30 seconds at 24 months after 1 or several ablation procedures with or without antiarrhythmic drugs
Arrhythmia Burden | From 3 months (blanking period) to 12 months and 24 months after the first ablation procedure
  Number of Registrations with Remote Heart Monitor / Number of Registrations with Atrial Arrhythmia with Remote Heart Monitor
Time to First Recurrens | From first ablation procedure to 24 months
  Time from first ablation procedure to first documented recurrens of atrial arrhythmias
Number of Repeat Procedures | 12 and 24 months after the first ablation procedure
  Number of repeat procedures
Changes in Quality of Life Measures: Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Overall Score and Subscale Scores | Baseline, 12 and 24 months after the first ablation procedure
  AFEQT is a 21 questions atrial fibrillation specific health related quality of life questionnaire. Overall Score (calculated from 18 of the questions) and subscale scores in three domains: symptoms, daily activities, and treatment concern. Score ranges from 0 to 100 points. Higher scores mean a better outcome.
Changes in Quality of Life Measures: RAND 36 (Research ANd Development) 36 All Domains | Baseline,12 and 24 months after the first ablation procedure
  RAND 36 (developed by RAND corporation) is a 36 questions health related quality of life questionnaire. The RAND 36 is divided into 8 domains: Physical functioning, role physical, role emotional, bodily pain, vitality, general health, social functioning and mental health. Score range from 0 to 100 points. Higher scores mean a better outcome.
Number of Participants with Adverse Events/ Complications | 12 and 24 months after the first ablation procedure
  Complications related to the ablation procedure: Cardiac perforation, stroke, transitory ischemic attack (TIA), systemic embolic events, atrio-esophageal fistula, major bleeding, atrioventricular block, groin hematoma requiring vascular surgery or extended hospitalization.
Number of Participants With All-cause Mortality | 12 and 24 months after the first ablation procedure
  Number of Participants With All-cause Mortality
Procedure time | Immediately after the procedure
  Time from start of groin punction to withdrawal of the catheters
Fluoroscopy time | Immediately after the procedure
  Total fluoroscopy time during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mats Jensen-Urstad, MD, Study Director — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Cosedis Nielsen J, Curtis AB, Davies DW, Day JD, d'Avila A, Natasja de Groot NMS, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T; Document Reviewers:. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Europace. 2018 Jan 1;20(1):e1-e160. doi: 10.1093/europace/eux274. No abstract available. PMID 29016840
- [Background] Tilz RR, Rillig A, Thum AM, Arya A, Wohlmuth P, Metzner A, Mathew S, Yoshiga Y, Wissner E, Kuck KH, Ouyang F. Catheter ablation of long-standing persistent atrial fibrillation: 5-year outcomes of the Hamburg Sequential Ablation Strategy. J Am Coll Cardiol. 2012 Nov 6;60(19):1921-9. doi: 10.1016/j.jacc.2012.04.060. Epub 2012 Oct 10. PMID 23062545
- [Background] Scherr D, Khairy P, Miyazaki S, Aurillac-Lavignolle V, Pascale P, Wilton SB, Ramoul K, Komatsu Y, Roten L, Jadidi A, Linton N, Pedersen M, Daly M, O'Neill M, Knecht S, Weerasooriya R, Rostock T, Manninger M, Cochet H, Shah AJ, Yeim S, Denis A, Derval N, Hocini M, Sacher F, Haissaguerre M, Jais P. Five-year outcome of catheter ablation of persistent atrial fibrillation using termination of atrial fibrillation as a procedural endpoint. Circ Arrhythm Electrophysiol. 2015 Feb;8(1):18-24. doi: 10.1161/CIRCEP.114.001943. Epub 2014 Dec 20. PMID 25528745
- [Background] Verma A, Wazni OM, Marrouche NF, Martin DO, Kilicaslan F, Minor S, Schweikert RA, Saliba W, Cummings J, Burkhardt JD, Bhargava M, Belden WA, Abdul-Karim A, Natale A. Pre-existent left atrial scarring in patients undergoing pulmonary vein antrum isolation: an independent predictor of procedural failure. J Am Coll Cardiol. 2005 Jan 18;45(2):285-92. doi: 10.1016/j.jacc.2004.10.035. PMID 15653029
- [Background] Oakes RS, Badger TJ, Kholmovski EG, Akoum N, Burgon NS, Fish EN, Blauer JJ, Rao SN, DiBella EV, Segerson NM, Daccarett M, Windfelder J, McGann CJ, Parker D, MacLeod RS, Marrouche NF. Detection and quantification of left atrial structural remodeling with delayed-enhancement magnetic resonance imaging in patients with atrial fibrillation. Circulation. 2009 Apr 7;119(13):1758-67. doi: 10.1161/CIRCULATIONAHA.108.811877. Epub 2009 Mar 23. PMID 19307477
- [Background] Rolf S, Kircher S, Arya A, Eitel C, Sommer P, Richter S, Gaspar T, Bollmann A, Altmann D, Piedra C, Hindricks G, Piorkowski C. Tailored atrial substrate modification based on low-voltage areas in catheter ablation of atrial fibrillation. Circ Arrhythm Electrophysiol. 2014 Oct;7(5):825-33. doi: 10.1161/CIRCEP.113.001251. Epub 2014 Aug 23. PMID 25151631
- [Background] Yagishita A, Sparano D, Cakulev I, Gimbel JR, Phelan T, Mustafa H, De Oliveira S, Mackall J, Arruda M. Identification and electrophysiological characterization of early left atrial structural remodeling as a predictor for atrial fibrillation recurrence after pulmonary vein isolation. J Cardiovasc Electrophysiol. 2017 Jun;28(6):642-650. doi: 10.1111/jce.13211. Epub 2017 May 29. PMID 28387462
- [Background] Schreiber D, Rieger A, Moser F, Kottkamp H. Catheter ablation of atrial fibrillation with box isolation of fibrotic areas: Lessons on fibrosis distribution and extent, clinical characteristics, and their impact on long-term outcome. J Cardiovasc Electrophysiol. 2017 Sep;28(9):971-983. doi: 10.1111/jce.13278. Epub 2017 Jul 5. PMID 28635186
- [Background] Kottkamp H, Bender R, Berg J. Catheter ablation of atrial fibrillation: how to modify the substrate? J Am Coll Cardiol. 2015 Jan 20;65(2):196-206. doi: 10.1016/j.jacc.2014.10.034. PMID 25593061
- [Background] Phlips T, Taghji P, El Haddad M, Wolf M, Knecht S, Vandekerckhove Y, Tavernier R, Duytschaever M. Improving procedural and one-year outcome after contact force-guided pulmonary vein isolation: the role of interlesion distance, ablation index, and contact force variability in the 'CLOSE'-protocol. Europace. 2018 Nov 1;20(FI_3):f419-f427. doi: 10.1093/europace/eux376. PMID 29315411
- [Background] El Haddad M, Taghji P, Phlips T, Wolf M, Demolder A, Choudhury R, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Determinants of Acute and Late Pulmonary Vein Reconnection in Contact Force-Guided Pulmonary Vein Isolation: Identifying the Weakest Link in the Ablation Chain. Circ Arrhythm Electrophysiol. 2017 Apr;10(4):e004867. doi: 10.1161/CIRCEP.116.004867. PMID 28381417